CLINICAL TRIAL: NCT07166757
Title: A Phase I/II Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of Human Allogeneic Induced Pluripotent Stem Cell-derived Dopaminergic Neural Progenitor Cell Injection in the Treatment of Early-onset Parkinson's Disease
Brief Title: Clinical Study to Evaluate XS411 in Treatment of Early-onset Parkinson's Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: XellSmart Bio-Pharmaceutical (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: XS411-Allo-EOPD-CN1/2-P01
Record Dates: First submitted 2025-08-06; First posted 2025-09-10 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease (PD)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 9.0×10^6 cells / bilateral putamen (Experimental)
  Interventions: Drug: human allogeneic induced pluripotent stem cell (iPSC)-derived dopaminergic neural progenitor cell injection
- 1.8×10^7 cells / bilateral putamen (Experimental)
  Interventions: Drug: human allogeneic induced pluripotent stem cell (iPSC)-derived dopaminergic neural progenitor cell injection

INTERVENTIONS:
Drug: human allogeneic induced pluripotent stem cell (iPSC)-derived dopaminergic neural progenitor cell injection — 5.0×10^7 cells/mL, injection, once, 12 months

SUMMARY:
This study is a Phase I/II clinical study to evaluate the safety, tolerability, and efficacy of XS411 in the treatment of EOPD. The study consists of two phases: Phase I and Phase II.

Phase I study is planned to be conducted in patients with EOPD, using a single-arm, open-label, traditional " 3+3 " dose-escalation design, aiming to investigate the safety, tolerability and preliminary efficacy of XS411 in the treatment of EOPD and to determine the RP2D.

Phase I study enrolls 6-12 patients with EOPD. Two dose cohorts (3-6 patients/dose cohort) are planned: 9×10⁶ cells /patient and 1.8 ×10⁷ cells /patient. Each participant will receive a single injection of XS411. Each participant in each dose cohort will be observed for at least 28 days after dosing . If no DLTs occur and the investigator has no other safety concerns for that participant, the next participant in that dose cohort will be enrolled.

Phase II study is planned for patients with EOPD, using a randomized, double-blind, sham-controlled, parallel-group design . The study will investigate the efficacy and safety of XS411 in the treatment of EOPD . Phase II study currently plans to enroll 81 patients with EOPD. The patients will be randomly assigned in a 2:1 ratio to either the experimental or control group. Participants in the experimental group will receive a single injection of XS411 in combination with an immunosuppressant at the RP2D determined during the Phase I dose-escalation phase (which may be adjusted based on the Phase II study results). The control group will receive a sham procedure in combination with an immunosuppressant sham.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤ age of onset ≤ 50 years old, diagnosed with EOPD (meeting the MDS 2015 clinical diagnostic criteria for Parkinson's disease );
* 18 years old ≤ age at enrollment ≤ 70 years old , male/female;
* Disease duration ≥ 5 years;
* Phase I: the modified Hoehn-Yahr grade in the off-phase is 3-4 (including the critical value) , and the modified Hoehn-Yahr grade in the on-phase is ≤3 ; Phase II: the modified Hoehn-Yahr grade in the off-phase is 2-4 (including the critical value) , and the modified Hoehn-Yahr grade in the on-phase is ≤3;
* Off-period MDS -UPDRS-III score >30;
* Positive L-dopa stress test;
* The patient is unable to adequately control motor fluctuations even with a stable dose of medication recommended in the "Guidelines for the Treatment of Parkinson's Disease in China (Fourth Edition)" ;
* Patients received stable doses of anti-PD drugs for at least 4 weeks before administration;
* Able to accept surgical anesthesia, suitable for neurosurgery under anesthesia, and able to undergo brain CT /MRI examination;
* Participants agree to postpone any other elective neurosurgery until the completion of the 24-month follow-up study;
* Participants agreed not to participate in any other clinical studies within 24 months after dosing;
* Participants or their legal representatives understand and comply with the research procedures, voluntarily participate and sign the ICF

Exclusion Criteria:

* Non-primary PD or Parkinson's superimposed syndromes ;
* Patients are in the late stages of PD and are experiencing severe, disabling peak-dose dyskinesia or biphasic dyskinesia and/or unpredictable or widely fluctuating symptoms;
* Have previously undergone neuronucleotomy, deep brain stimulation (DBS), striatal surgery, extrapyramidal surgery, stereotactic brain surgery, or other brain surgery; or who have undergone other surgical procedures that the investigator determined would affect participation in this study; or who have surgical contraindications
* Patients currently receiving L-dopa intestinal instillation, apomorphine injection, or continuous daily infusion of anti-PD drugs;
* Patients who had used botulinum toxin, phenol, subarachnoid injection of baclofen, or received interventional treatment for dystonia or spasticity within 6 months before medication;
* Have used glucocorticoids or immunosuppressive drugs for a long time within 3 months before the screening visit;
* Those who have received cell therapy before;
* Patients who received electroconvulsive therapy within 30 days before administration;
* Those who have received or plan to receive vaccines during the trial within 3 months before screening, such as vaccines for novel coronavirus pneumonia (COVID-19), influenza, herpes zoster, and pneumococcal vaccine;
* Those with a history of mental illness who are judged by the researchers to be unsuitable for study participation; or those with severe suicidal ideation currently or within the year before screening or any history of suicide attempts within the past 2 years;
* Those with active epilepsy or currently taking anti-epileptic drugs;
* Those with a history of dementia or severe cognitive impairment; or those with obvious dementia or cognitive impairment at screening; dementia may affect participants' poor compliance, inability to accurately record diaries, and / or inability to sign the ICF;
* Severe anxiety at screening;
* Patients whose previous head CT/MRI examinations showed brain injuries such as brain trauma, cerebral vascular malformation, hydrocephalus, brain tumors, or abnormal brain imaging of the striatum and other brain regions, which significantly increased the surgical risk;
* Those with uncontrolled autoimmune diseases;
* Patients with a history of severe cardiovascular and cerebrovascular diseases;
* Patients with other serious systemic diseases;
* During the screening period, patients have severe arthritis, limp, severe sequelae of stroke, severe osteoporosis, or a history of severe trauma within 1 month (such as hip or lower limb fractures), which may affect the study evaluation as assessed by the researchers;
* Patients with malignant tumors or a history of malignant tumors;
* Patients with active disseminated intravascular coagulation and obvious bleeding tendency within 3 months before signing the ICF, or patients who cannot stop taking antiplatelet drugs or other anticoagulants for at least 10 days before surgery;
* Previous history of abnormal coagulation function;
* Patients with lab result abnormalities during screening include;
* Allergic to the drugs used in the study;
* Are pregnant or breastfeeding, or plan to become pregnant during the study;
* Female participants of fertile potential must have a positive pregnancy test result before dosing; female participants of fertile potential, or male participants who are not sterilized and whose partners are fertile, must not take effective contraceptive measures from the time they sign the ICF until at least 24 months after dosing; female participants must not agree to not donate eggs from the time they sign the ICF until at least 24 months after dosing, and male participants must not agree to not donate sperm from the time they sign the ICF until at least 24 months after dosing;
* Participants who are currently participating in other clinical trials, or have participated in other clinical studies and received intervention treatment within 1 month before administration;
* Those who are considered by the researchers to have poor compliance;
* Any other situation that the researcher deems to jeopardize the safety of the participants or affect the study evaluation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of XS411 cell injection in the treatment of EOPD 28 days after administration | 28 days after treatment
  To evaluate the safety and tolerability of XS411 cell injection in the treatment of EOPD through the incidence and severity of AEs/SAEs; the incidence of DLTs ; Vital signs, physical examination, 12-lead ECG, clinical laboratory tests, and head MRI.
  AEs occurring during the study will be graded according to CTCAE V5.0. DLT is defined as: (1) any CTCAE grade 3 or 4 AE related to the trial drug (including definitely related, probably related, and possibly related) occurring within 28 days of trial drug administration (such as grade 3 or 4 immune system diseases, infectious diseases, mental illnesses, kidney diseases, etc. related to the trial drug ); (2) Grade 2 AEs cannot be reduced to grade 1 or below within 14 days.

SECONDARY OUTCOMES:
To check the change on parameters in MDS-UPDRS questionnaire on Day 28, M3, M6, M9 and M12 to evaluate preliminary efficacy of XS411 cell injection. | 28 days, 3, 6, 9, and 12 months after administration
  To evaluate the preliminary efficacy of XS411 cell injection in the treatment of EOPD through Changes from baseline in the scores of parts I, II, III, and IV of the MDS-UPDRS (individual scores, total score, and sum of scores II and III) after administration ;
Evaluation of the improvement of nigrostriatal dopamine transmitter system through PET-CT testing data change compared with baseline in M6 and M12 for 9 partipants | 6 and 12 months after administration
  To evaluation of the improvement of nigrostriatal dopamine transmitter system after XS411 cell injection in the treatment of EOPD through 18F-DOPA uptake in the striatum as shown by brain PET-CT at 6 and 12 months after administration compared with baseline.
To check the change on parameters Hoehn-Yahr (modified) questionnaire on Day 28, M3, M6, M9 and M12 to evaluate preliminary efficacy of XS411 cell injection. | 28 days, 3, 6, 9, and 12 months after administration
  To evaluate the preliminary efficacy of XS411 cell injection in the treatment of EOPD through Change from baseline in the Hoehn-Yahr (modified) Parkinson's disease rating scale score after administration ;
To check the change on parameters on OFF and ON-period change recorded in patient's diary on Day 28, M3, M6, M9 and M12 to evaluate preliminary efficacy of XS411 cell injection. | 28 days, 3, 6, 9, and 12 months after administration
  To evaluate the preliminary efficacy of XS411 cell injection in the treatment of EOPD through Change from baseline in on-period without bothersome dyskinesia; Change from baseline in conscious off-period; Change from baseline in on-period without dyskinesia recorded in Patient's diary

OTHER OUTCOMES:
Evaluation of the improvement of nigrostriatal dopamine transmitter system after XS411 cell injection in the treatment of EOPD | 6 and 12 months after administration
  To evaluation of the improvement of nigrostriatal dopamine transmitter system after XS411 cell injection in the treatment of EOPD through PET-CT testing data change compared with baseline in M6 and M12 for 9 partipants in the striatum as shown by brain PET at 6 and 12 months after administration compared with baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes